CLINICAL TRIAL: NCT00560625
Title: Low Dose(1mcg) ACTH Stimulation Test for Assessment of the Hypothalamus-pituitary-adrenal Axis in Patients Treated With Inhaled Busedonide or Fluticasone.
Brief Title: Does Inhaled Busedonide or Fluticasone Impair Adrenal Function?
Status: Terminated | Type: Observational
Why Stopped: recruiting subjects did not start.
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 0030-07EMC
Record Dates: First submitted 2007-11-18; First posted 2007-11-20 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Inhaled corticosteroids are largely used in patients with asthma or chronic obstructive lung diseases. The purpose of this study is to determine if the use of inhaled corticosteroids is associated with suppression of endogenous cortisol production, as seen in patients treated with pharmacologic doses of oral or parenteral steroids.

DETAILED DESCRIPTION:
The normalcy of the hypothalmic-pituitary-adrenal (HPA) axis of enrolled subjects will be assessed by low dose (1mcg) corticotropin (ACTH)stimulation test. Serum cortisol levels will be measured before , 30 minutes and 60 minutes after 1 mcg ACTH intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving inhaled busedonide or fluticasone at daily dose of 200-800 mcg ' for at least 4 weeks

Exclusion Criteria:

* patients receiving any corticosteroid therapy, except inhaled busedonide or fluticasone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital-based respiratory diseases clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
stimulated serum cortisol levels | within 30 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Ishay, MD, Principal Investigator — Endocrine Institute , Haemek Medical Center, Afula. 18101 Israel
Locations (1):
- Endocrine Institute, Haemek medical Center, Afula, Israel